CLINICAL TRIAL: NCT02394431
Title: Added Value of Speckle Tracking in the Evaluation of Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Marielle Morissens, Deputy Head of Clinic, Brugmann University Hospital
Other Study IDs: CHUB-Echo-Cardio
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Echocardiography; Speckle tracking
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sickle cell disease patients: Sickle cell disease patients
  Interventions: Other: Cardiac echography; Other: Biological parameters; Other: Clinical parameters
- Healthy patients: This is the control group for the sickle cell disease patients: each sickle cell disease patient will be matched with a healthy patient of the same sex and of similar age.
  Interventions: Other: Cardiac echography; Other: Biological parameters

INTERVENTIONS:
Other: Cardiac echography — Ejection fraction measured by Teicholz and planimetry, diastolic function, tissular doppler, myocardiac performance index, global longitudinal strain measured by speckle tracking, arterial pulmonary hypertension, left ventricular hypertrophy.
Other: Biological parameters — Hemoglobin levels, red cells, hematocrit, iron, ferritin
Other: Clinical parameters — Blood transfusion number, severity of the sickle cell disease damage, evolution duration of the sickness
  Groups: Sickle cell disease patients

SUMMARY:
Sickle Cell Disease is a serious disease that is life-threatening for patients being homozygous for the SS form or heterozygous for the SC or βthal forms. The CHU Brugmann hospital currently regularly treats about 70 homozygous adult patients and this number is in constant augmentation.

Sickle cell disease patients may develop a cardiomyopathy due to chronic anemia, the haemosiderosis risk or, less frequently, to coronary vaso-occlusive damages.

The hypervolemia in patients with sickle cell disease causes an overestimation of the ejected left ventricular fraction measured by echocardiography, this parameter being very dependent of the blood volume.It has already been shown that the left ventricular ejection fraction was normal in most patients with sickle cell disease, but that its evaluation by parameters independent from the blood volume showed the existence of a dysfunction.

Myocardial strain, as measured by speckle tracking, is a echographic evaluation method of the cardiac function, independent of the blood volume. This technique hasn't been used much in sickle cell disease patients. A study using 3D speckle tracking on a limited number of sickle cell disease patients failed to show a strain anomaly. Moreover, the study highlighted a higher global longitudinal strain in this patient population. The investigators find these data hard to explain and in contradiction with previous studies using other cardiac function evaluation techniques, independent from the blood volume.

The primary goal of this study is thus

* to study the longitudinal strain by 2D echography
* to determine if anomalies of the longitudinal strain exist in sickle cell disease patients with a normal ejected left ventricular fraction, compared to a control group of healthy patients.

The secondary goal of this study is to correlate, inside the sickle cell disease group, the possible strain anomalies with biological gravity parameters of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All sickle cell disease patients

Exclusion Criteria:

* Insufficient echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sickle cell disease patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cardiac ejection fraction | once per year, at the annual medical visit planned according to the standart of care for this pathology
  Ejection fraction measured by Teicholz and planimety.
Cardiac diastolic function | once per year, at the annual medical visit planned according to the standart of care for this pathology
Cardiac tissular doppler | once per year, at the annual medical visit planned according to the standart of care for this pathology
Myocardiac performance index | once per year, at the annual medical visit planned according to the standart of care for this pathology
Global longitudinal strain | once per year, at the annual medical visit planned according to the standart of care for this pathology
  Global longitudinal strain measured by speckle tracking.
arterial pulmonary hypertension | once per year, at the annual medical visit planned according to the standart of care for this pathology
left ventricular hypertrophy | once per year, at the annual medical visit planned according to the standart of care for this pathology

SECONDARY OUTCOMES:
Biological parameters: hemoglobin levels | once per year, at the annual medical visit planned according to the standart of care for this pathology
Biological parameters: ferritin levels | once per year, at the annual medical visit planned according to the standart of care for this pathology
Biological parameters: red cells count | once per year, at the annual medical visit planned according to the standart of care for this pathology
Biological parameters: hematocrit levels | once per year, at the annual medical visit planned according to the standart of care for this pathology
Biological parameters: iron levels | once per year, at the annual medical visit planned according to the standart of care for this pathology
Clinical parameters: severity of the illness | once per year, at the annual medical visit planned according to the standart of care for this pathology
  Sickle cell disease organ damages.
Clinical parameters: sanguine transfusion numbers | once per year, at the annual medical visit planned according to the standart of care for this pathology

CONTACTS AND LOCATIONS:
Overall Officials: Marielle MORISSENS, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Ahmad H, Gayat E, Yodwut C, Abduch MC, Patel AR, Weinert L, Desai A, Tsang W, Garcia JG, Lang RM, Mor-Avi V. Evaluation of myocardial deformation in patients with sickle cell disease and preserved ejection fraction using three-dimensional speckle tracking echocardiography. Echocardiography. 2012 Sep;29(8):962-9. doi: 10.1111/j.1540-8175.2012.01710.x. Epub 2012 May 8. PMID 22563937
- [Background] Knight-Perry JE, de las Fuentes L, Waggoner AD, Hoffmann RG, Blinder MA, Davila-Roman VG, Field JJ. Abnormalities in cardiac structure and function in adults with sickle cell disease are not associated with pulmonary hypertension. J Am Soc Echocardiogr. 2011 Nov;24(11):1285-90. doi: 10.1016/j.echo.2011.07.009. Epub 2011 Aug 27. PMID 21873028
- [Background] Sachdev V, Machado RF, Shizukuda Y, Rao YN, Sidenko S, Ernst I, St Peter M, Coles WA, Rosing DR, Blackwelder WC, Castro O, Kato GJ, Gladwin MT. Diastolic dysfunction is an independent risk factor for death in patients with sickle cell disease. J Am Coll Cardiol. 2007 Jan 30;49(4):472-9. doi: 10.1016/j.jacc.2006.09.038. Epub 2007 Jan 16. PMID 17258093
- [Background] Hankins JS, McCarville MB, Hillenbrand CM, Loeffler RB, Ware RE, Song R, Smeltzer MP, Joshi V. Ventricular diastolic dysfunction in sickle cell anemia is common but not associated with myocardial iron deposition. Pediatr Blood Cancer. 2010 Sep;55(3):495-500. doi: 10.1002/pbc.22587. PMID 20658621
- [Background] Voskaridou E, Christoulas D, Terpos E. Sickle-cell disease and the heart: review of the current literature. Br J Haematol. 2012 Jun;157(6):664-73. doi: 10.1111/j.1365-2141.2012.09143.x. Epub 2012 Apr 25. PMID 22530942
- [Background] Poludasu S, Ramkissoon K, Salciccioli L, Kamran H, Lazar JM. Left ventricular systolic function in sickle cell anemia: a meta-analysis. J Card Fail. 2013 May;19(5):333-41. doi: 10.1016/j.cardfail.2013.03.009. PMID 23663816